

Doc Number: 104-09200

**Revision: A** 

# **ACHIEVE GRX Registry Summary**

TITLE A Post-Market Registry for the Evaluation of the CorPath®

GRX System Effectiveness in Peripheral Vascular Interven-

tions

SHORT TITLE: ACHIEVE GRX Registry

**DEVICE** CorPath GRX System:

 The Bedside Components consist of an Extended Reach Arm, Robotic Drive and Single-use Cassette

• Interventional Cockpit

• Control Console

**REGULATORY STATUS** The CorPath GRX was granted 510K clearance (K173288) for

use in peripheral interventions on February 15, 2018, and was

CE Marked effective March 07, 2018 (CE 549879).

**INDICATION FOR USE** The CorPath GRX System is intended for use in the remote

delivery and manipulation of guidewires and rapid exchange catheters, and remote manipulation of guide catheters during

percutaneous coronary and vascular procedures.

**STUDY OBJECTIVE** To collect data on the routine patterns of use, safety and effec-

tiveness, including the clinical and technical performance of the CorPath GRX System, in the delivery and manipulation of guidewires and rapid exchange catheters and manipulation of guide catheters during peripheral vascular intervention (PVI)

procedures.

STUDY DESIGN This is a prospective, single-arm, open-label, multi-center pa-

tient registry of the CorPath GRX System to examine its performance during peripheral vascular interventions and patient outcomes through 24 hours post-procedure or hospital dis-

charge, whichever occurs first.

CO-PRINCIPAL Dr. Jon George

**INVESTIGATORS** Einstein Medical Center

5501 Old York Road Philadelphia, PA 19141

Dr. John Phillips

Riverside Methodist Hospital

3705 Olentangy River Rd, Suite 100

Columbus, OH 43214

**SAMPLE SIZE** It is expected that up to 200 subjects shall be enrolled in the

study.



Doc Number: 104-09200

**Revision: A** 

#### **EVALUATION PERIOD**

Estimated date of first patient enrolled: October 2020

Anticipated enrollment period: 24 months

Estimated date of last patient enrolled: October 2022

# INVESTIGATIONAL SITES

It is expected that up to 10 centers (USA and International) may participate in this study.

# STUDY DURATION/ FOLLOW-UP PERIOD

All subjects will be followed post-CorPath percutaneous vascular intervention through 24 hours post-procedure or hospital discharge, whichever occurs first.

# SUBJECT POPULATION

Subjects with a clinical indication for Peripheral Vascular Intervention (PVI).

## PATIENT GENERAL IN-CLUSION CRITERIA

Candidates will be included in the study only if all the following conditions are met:

- 1. Age ≥ 18 years.
- 2. Subject has a clinical indication for Peripheral Vascular Intervention (PVI).
- 3. Subject is deemed appropriate for robotic-assisted PVI.
- 4. The subject has been informed of the nature of the study, agrees to its provisions and has provided written informed consent.
- 5. Individual monitoring of radiation dose, using the pocket dosimeter, was initiated at start of procedure.

# PATIENT GENERAL EX-CLUSION CRITERIA

Candidates will be excluded from the study if any of the following conditions are present:

- 1. Failure/inability/unwillingness to provide informed con-
- 2. The investigator determines the subject or the peripheral anatomy is not suitable for robotic-assisted PVI.
- 3. Women who are pregnant.

## STAFF GENERAL IN-CLUSION CRITERIA

Staff members may participate in the study only if all the following conditions are met:

- 1. Interventional lab staff, including the operating physician, secondary operator, and, if applicable, ancillary staff (technician and nurse).
- 2. Interventional lab staff member has been informed of the nature of the study, agrees to its provisions, and has provided written informed consent.

## STAFF GENERAL EX-CLUSION CRITERIA

Staff members will be excluded from the study if any of the following conditions are present:



Doc Number: 104-09200

**Revision: A** 

 Failure/inability/unwillingness to provide informed consent

- Interventional lab staff members who are undergoing medical treatment involving additional radiation exposure
- 3. Interventional lab staff members who have exceeded their hospital defined dose limits for radiation anytime during their participation in the study.

# PRIMARY EFFECTIVENESS END-POINT

#### **Technical Success**

The primary effectiveness endpoint will be defined as successful completion of the robotic-assisted endovascular procedure absent any unplanned conversion to manual for guidewire or balloon/stent catheter inability to navigate vessel anatomy.

#### Clinical Success

Defined as <30% residual stenosis in all CorPath GRX System treated lesions at the completion of the interventional procedure in the absence of device-related serious adverse events (SAE), either within twenty-four (24) hours of the procedure or prior to hospital discharge, whichever occurs first.

## PRIMARY SAFETY ENDPOINT

The primary safety endpoint will be a composite of intra- and peri-procedural events, including target vessel rupture, clinically significant perforation or dissection, and distal embolization, within 24-hours post-procedure or hospital discharge, whichever occurs first.

# SECONDARY ENDPOINTS

#### **PVI Procedure Time**

Defined as the time measured from the insertion of the guiding sheath until the removal of the guiding sheath.

#### Manual time

Defined as the total amount of time the procedure is completed using a manual technique.

#### **Robotic Time**

Defined as the total amount of time the procedure is completed robotically from the robotic cockpit.

#### Fluoroscopy Time

Total fluoroscopy utilized during the procedure as recorded by an Imaging System.



Doc Number: 104-09200

**Revision: A** 

## **Operator Radiation Exposure**

Cumulative dose the operator receives as recorded from an electronic pocket dosimeter during the procedure.

## **Staff Radiation Exposure**

Cumulative dose the staff receives as recorded from an electronic pocket dosimeter during the procedure.

## **Patient Radiation Exposure**

DAP (dose-area-product) and AK (air kerma) as recorded during the procedure.

### **Contrast Fluid Volume**

Total volume of contrast (mL) used during the procedure.

STUDY SPONSOR Corindus, Inc.

309 Waverley Oaks Road, Suite 105

Waltham, MA 02452 USA

MANUFACTURER Corindus, Inc.

309 Waverley Oaks Road, Suite 105

Waltham, MA 02452 USA

MONITORING Corindus, Inc.

**SERVICE** 309 Waverley Oaks Road, Suite 105

Waltham, MA 02452 USA

**DATA** MedNet Solutions, Inc.

**COORDINATING** 110 Cheshire Lane, Suite 300 **CENTER** Minnetonka, MN 55305 USA

**STATISTICAL** Technomics Research ANALYSIS 1815 Medina Road

SERVICES Long Lake, MN 55356 USA